CLINICAL TRIAL: NCT00136227
Title: Trial of Interventions to Increase Utilization of Colorectal Cancer Screening and Promote Informed Decision Making About Colorectal Cancer Screening Among Hispanic Men and Women
Brief Title: Use and Decision-making About Colorectal Cancer Screening Among Hispanic Men and Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCCDPHP-4527; U48/DP000057 (SIP 18-04); U48DP000057 (NIH)
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Last update posted 2012-09-07 (Estimated); Status verified 2012-09

CONDITIONS: Colorectal Cancer
Keywords: screening,; community health education,; decision making,; computer-assisted decision making
MeSH Terms: conditions — Colorectal Neoplasms; Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lifestyle counseling (Experimental): Behavioral: small media intervention using video, flip chart, and pamphlets and a tailored interactive multimedia intervention
  Interventions: Behavioral: small media intervention using video, flip chart, and pamphlets and a tailored interactive multimedia intervention

INTERVENTIONS:
Behavioral: small media intervention using video, flip chart, and pamphlets and a tailored interactive multimedia intervention

SUMMARY:
During this first year, the researchers have worked toward identifying factors influencing initiation of colorectal cancer screening among Hispanic men and women aged 50 and older and developing an intervention plan using Intervention Mapping, a framework for systematic health promotion program planning, implementation, and evaluation. The researchers are also currently in the preliminary stages of developing two promotora (lay health worker)-delivered interventions: a small media intervention (video, flip chart, pamphlets) and a tailored interactive multimedia intervention, prior to the actual collection of data. Thus, although 733 subjects have been approved by the Committee for the Protection of Human Subjects to be enrolled in this study in the future, no subjects have been enrolled at this time. Consequently, there have been no adverse events, and since the risks associated with participating in this study are negligible, the researchers do not anticipate any adverse events in the future. No modifications have been made to the research since the last review, other than that the researchers are currently reassessing the need to conduct preliminary qualitative research as proposed in the original protocol.

DETAILED DESCRIPTION:
During this first year, the researchers have worked toward identifying factors influencing initiation of colorectal cancer screening among Hispanic men and women aged 50 and older and developing an intervention plan using Intervention Mapping, a framework for systematic health promotion program planning, implementation, and evaluation. The researchers are also currently in the preliminary stages of developing two promotora (lay health worker)-delivered interventions: a small media intervention (video, flip chart, pamphlets) and a tailored interactive multimedia intervention, prior to the actual collection of data. Thus, although 733 subjects have been approved by the Committee for the Protection of Human Subjects to be enrolled in this study in the future, no subjects have been enrolled at this time. Consequently, there have been no adverse events, and since the risks associated with participating in this study are negligible, the researchers do not anticipate any adverse events in the future. No modifications have been made to the research since the last review, other than that the researchers are currently reassessing the need to conduct preliminary qualitative research as proposed in the original protocol.

ELIGIBILITY:
Exclusion Criteria:

* Personal history of colorectal cancer

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 521 (Actual)
Dates: Start 2005-10; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
colorectal cancer screening initiation rate | 30 days

SECONDARY OUTCOMES:
decisional balance | 30 days
self-efficacy | 30 days
knowledge about colorectal cancer screening | 30 days
perceived risk of colorectal cancer | 30 days
perceived survivability | 30 days
perceived guilt | 30 days
outcome expectations | 30 days
subjective norms | 30 days
intention to undergo colorectal cancer screening | 30 days
making decisions about colorectal cancer screening that are consistent with their values and preferences | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Maria E. Fernandez, PhD, Principal Investigator — University of Texas at Houston
Locations (1):
- University of Texas, Houston, Texas, United States